CLINICAL TRIAL: NCT01885598
Title: Eliquis (Apixaban) Regulatory Postmarketing Surveillance in Clinical Practice for Stroke Prevention in Nonvalvular Atrial Fibrillation
Brief Title: Eliquis Regulatory Post Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-259
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: NonValvular Atrial Fibrillation
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nonvalvular Atrial Fibrillation patients with risk of Stroke: Patients undergoing elective total hip replacement arthroplasty or elective total knee replacement arthroplasty and signed on the data release
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis

SUMMARY:
The primary objective of this study is to examine the safety profile of Eliquis in Korean nonvalvular atrial fibrillation patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients ≥19 years of age
* Adult patients who are diagnosed with nonvalvular atrial fibrillation and are initiating Eliquis anticoagulation therapy for risk reduction of stroke and systemic embolism
* Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Receiving Eliquis treatment for an indication that is not approved in Korea
* Contraindicated for the use of Eliquis as described in the Korean label

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting outpatient department of hospital
Sampling Method: Non-Probability Sample
Enrollment: 3335 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) occurrence based on Incidence of serious adverse events, unexpected adverse drug reactions, Identification of AE profile in usual practice Nonserious adverse events, major bleeding | within 30 days after end of the treatment

SECONDARY OUTCOMES:
Final identification of major events and no event based on Incidence of stroke, systemic embolism, death, Effectiveness or death at 24 months after discontinuation of therapy or at the end of the observation period (whatever is later) | At 3, 6, 12, and 24 months after enrollment
  Final identification of major events based on Incidence of stroke, systemic embolism, death, Effectiveness: No evidence of stroke, systemic embolism, or death at 24 months after discontinuation of therapy or at the end of the observation period (whatever is later)
Final evaluation of clinical significance of Eliquis is provided by the physician's subjective decision (Excellent, Good, Moderate, Insufficient) | At 3, 6, 12, and 24 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- [Derived] Kim JS, Koo J, Shin DI, Kim BS, Kim J, Kim EG, Hong KS, Yi H. Apixaban for Secondary Stroke Prevention: Coexistant Cerebral Atherosclerosis May Increase Recurrent Strokes. J Stroke. 2022 Jan;24(1):118-127. doi: 10.5853/jos.2021.02355. Epub 2022 Jan 31. PMID 35135065
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx